CLINICAL TRIAL: NCT04614870
Title: Non-interventional, Prospective, Single-blinded, Observational, Multicenter, Cohort, Clinical Study to Evaluate DETEC® Esterase for the Detection of Infections in Chronic Wounds
Brief Title: DETEC® Esterase for Screening Wound Infection at Point of Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Progenitec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DETEC 002
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: DETEC® Esterase — DETEC® Esterase is a disposable diagnostic device that is used to indicate the presence or absence of infection based on the presence or absence of the evaluated level of leukocyte esterase by testing the freshly recovered wound dressing which are soaked with wound exudate.

SUMMARY:
This non-interventional, single-blinded, prospective, observational study assesses the planar distribution of leukocyte esterase in wounds by placing wound exudates soaked wound dressings in the DETEC® Esterase device during routine wound care. The output of the device is correlated with clinical determination of infection to assess the device efficacy in identifying presumptive infections.

DETAILED DESCRIPTION:
There is no commercial available device to diagnosze infection in chronic wounds. Since qualitative measures of leukocyte esterase (LE) have been used clinically as a biomarker to screen for various infectious diseases including urinary tract infections, peritonitis and joint infections, it is likely that LE can also be used a a biomarker to screen infection in chronic wounds. To test this hypothesis, an investigational device - DETEC® Esterase - has been developed to detect elevated LE in wound exudates absorbed wound dressings. With increasing LE levels, this coloration becomes more intense (from colorless/pink to dark purple) indicating infection.

The overall goals of the study are as follows:

1. To assess the efficacy of DETEC® Esterase in detecting ulcer wound infection by comparing device output with the wound care specialist's final determination of infection
2. To evaluate the effect of the subject's age, race, wound size, location, type, and clinical site on the device's ability to identify non-healing wounds.
3. To study the sensitivity, specificity, and accuracy of DETEC® Esterase in assessing infection by testing discarded wound dressings with varying levels of esterase activities.

Patients presenting themselves to the clinic with ulcer wounds will be assessed by the clinicians. Those with at least one clinical sign and symptom of a wound infection will be enrolled and recorded in the study. The participant's first visit can be concurrent with enrollment. During this visit, the participants' wound dressings will be tested using DETEC® Esterase device by a project nurse/tester not involved with subjects' wound management and the output recorded. Wounds will be managed by the clinicians who are blinded from the device output. Consequently, the clinician may adjudicate the presence or absence of infection based on all available information to make a clinical diagnosis of infection. The device determination of presumptive infection will then be compared with the results of the doctor's adjudication.

ELIGIBILITY:
Inclusion Criteria:

* Adult (21 years), male or female, inpatient/outpatient, presenting with a wound
* Chronic wound open for at least 30 days, including (Diabetic foot ulcers (DFU), Wagner grade 1 to 3), (Pressure ulcers, stage 2 to 4), (Venous leg ulcers (VLU), confirmed by venous duplex/Doppler),
* For wounds on a lower extremity (i.e. DFU, VLU) an ankle-brachial index (ABI) of greater than 0.6 for the affected leg to ensure ischemia will not impact healing
* For diabetic foot ulcers - confirmed type 1 or type 2 diabetes mellitus with a hemoglobin A1C less than 10 percentage
* Wound shows clinical signs of infection - pain, erythema, edema, heat, surrounding erythema, swelling, or purulent exudate

Exclusion Criteria:

* History of autoimmune disease/ acquired immunodeficiency syndrome/Hepatitis
* Require treatment for primary or metastatic malignancy
* Any contra-indication to routine wound care and/or monitoring
* Women who are pregnant, lactating, or of childbearing potential and currently not taking adequate birth control
* Participation (less than 30 days prior to baseline) in an interventional trial which could have a potential effect on the study outcome, as determined by the Investigator
* Patients with a dry dressing

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic wounds
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of the device in the determination of infection in wounds with clinical signs of infection | 15 days from enrollment
  The primary endpoint is agreement in infected wound determination between device output and providers' adjudication in wounds with suspected infection.

SECONDARY OUTCOMES:
Positive predictive value of the device in the determination of infection in wounds with various patient and wound conditions | 15 days from enrollment
  The secondary endpoint is identifying infection in wounds with various biometry and disease conditions (age, gender, race, wound size, wound locations, wound types, infection status, and clinical sites).
Likelihood of infection | 15 days from enrollment
  Another secondary endpoint is the likelihood of infection with positive and negative test results

CONTACTS AND LOCATIONS:
Overall Officials: Wenjing Hu, PhD, Principal Investigator — Progenitec Inc.
Locations (1):
- Complex Healthcare Solutions, Arlington, Texas, United States